CLINICAL TRIAL: NCT02363595
Title: Genomic Predictors of Papillary Microcarcinoma Disease Progression
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ohio State University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 14-277
Record Dates: First submitted 2015-02-05; First posted 2015-02-16 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Papillary Microcarcinoma
Keywords: Genomic Predictors; 14-277
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue

GROUPS / COHORTS (1):
- Papillary Microcarcinoma: This clinical trial protocol describes implementation of a prospective observation protocol to standardize data collection and obtain permission to collect samples of PMC tumors in a cohort of PMC patients being followed with active surveillance. This will allow PMC tumors to be accurately classified as either stable or progressive over time and used for comprehensive molecular profiling if surgical removal is required during follow-up

SUMMARY:
The study is being done to answer the following question: What are the specific clinical and molecular features that will help us predict which small thyroid cancers are likely to grow and be problematic?

Therefore, the purpose of this study is to identify specific clinical and molecular characteristics that are predictive of tumor progression in small thyroid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven papillary thyroid cancer (or suspicious for papillary thyroid cancer) confirmed by MSKCC cytopathologist.
* Being followed with active surveillance at MSKCC
* Biopsied index nodule less than or equal to 2 cm in maximum dimension
* Thyroid and neck US performed and interpreted by a MSKCC radiologist within 6 months prior to study entry.

Exclusion Criteria:

* Biopsied index nodule greater than 2 cm in any dimension
* Age less than 18 yrs old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All papillary thyroid cancer patients evaluated at MSKCC clinic.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
estimate the disease progression rate | 4 years
  Therefore, in order to ensure that we will have at least 459 patients with PTC being followed with active surveillance, we plan to enroll 500 total patients, of which 350 will have FNA diagnostic for PTC (of which 99% are expected to have PTC) and 150 patients will have FNA suspicious for PTC (of which 113 would be expected to have PTC). This sample size will enable us to estimate the 5 year disease progression rate requiring intervention to within ±4% at 95% confidence level (using binomial calculation under the assumption that the study is not stopped early and the progression rate is not higher than 10%).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tuttle, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/